CLINICAL TRIAL: NCT01016899
Title: Xoft Electronic Brachytherapy Clinical Protocol For The Primary Treatment Of Non-Melanoma Skin Cancer
Brief Title: Electronic Brachytherapy for the Treatment of NMSC
Status: Completed | Type: Observational
Sponsor: Xoft, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CTPR-0002
Record Dates: First submitted 2009-11-13; First posted 2009-11-20 (Estimated); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Basal Cell Carcinoma; Squamous Cell Carcinoma
Keywords: Electronic; Brachytherapy; Nonmelanoma; cancer
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Non-melanoma skin cancer: Early stage squamous or basal cell carcinoma
  Interventions: Radiation: electronic brachytherapy

INTERVENTIONS:
Radiation: electronic brachytherapy — Post market observational study recording data form patients with skin cancer treated with electronic brachytherapy. Treatment is standard of care, and can vary in dose and fractionation schedule from patient to patient depending on radiation oncologist's judgement for best treatment for the patient.
  Other Names: Xoft Axxent System

SUMMARY:
The objective of this study is to record recurrence in patients treated for nonmelanoma (basal cell and squamous cell carcinomas) skin cancer using the Xoft Axxent Electronic Brachytherapy System. Additional objectives include evaluate the appearance of the treated area in patients treated for nonmelanoma skin cancer using the Xoft Axxent Electronic Brachytherapy System and record the occurrence of radiation therapy related skin changes in patients treated for nonmelanoma skin cancer.

DETAILED DESCRIPTION:
The objective of this study is to record local recurrence in patients treated for nonmelanoma (basal cell and squamous cell carcinomas) skin cancer using the Xoft Axxent Electronic Brachytherapy System. Additional objectives include evaluate the cosmetic outcomes in patients treated for nonmelanoma skin cancer using the Xoft Axxent Electronic Brachytherapy System and record the occurrence of radiation therapy related skin toxicities in patients treated for nonmelanoma skin cancer using the Xoft Axxent Electronic Brachytherapy System.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed the informed consent form
* Pathological diagnosis confirmed of squamous cell or basal cell carcinoma
* Histopathological Grade: G1 (well differentiated), G2 (moderately differentiated), or Gx (Not assessed in report)
* Clinical Staging Tis, T1, or T2 (Must be ≤ 4 cm in diameter)
* One lesion is treated, or more than 1 lesion is treated with a minimum of a 5 mm gap between the edges of the lesion margins.

Exclusion Criteria:

* T2 > 4 cm and T3 and T4
* American Joint Committee Staging for NMSC Stages III and IV
* Histopathologic Grade 3 (poorly differentiated) or higher grade
* Target area is adjacent to a burn scar
* Target area is on the lip
* Patient < 50 years of age
* Any prior definitive surgical resection of the cancer
* Perineural invasion
* Lesion depth > 5mm on clinical assessment or as assessed by ultrasound or CT.
* Patient is pregnant (pregnancy test required if standard of care).
* Target area is prone to trauma.
* Target area with compromised lymphatic or vascular drainage.
* Participation in another investigational device or drug study concurrently.
* Patient has undergone prior radiation therapy to this specific anatomic location.
* Patient is receiving pharmacologic agent(s) at or around the time of the Radiation therapy that is/are known to produce skin reactions that will influence cosmesis grading during study.
* Patient is receiving chemotherapeutic agent(s) Six (6) weeks before or six (6) weeks after radiation therapy.
* Life expectancy less than five (5) years.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary basal cell and primary squamous cell carcinomas
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Local recurrence of NMSC | at six (6) months, one (1) year, two (2) years, three (3) years, four (4) years, and five (5) years.
  Local recurrence

SECONDARY OUTCOMES:
Cosmetic outcomes for patients treated for NMSC | (1) month, three (3) months, six (6) months, one (1) year, two (2) years, three (3) years, four (4) years, and five (5) years.
  Cosmetic outcomes
Occurrence of radiation therapy related skin toxicities | 1, 3, 6 months, and 1, 2, 3, 4, and 5 years
  Skin toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Bhatnagar, MD, MBA, Principal Investigator — Cancer Treatment Services-AZ
Locations (5):
- United States (5):
  - DCH Cancer Center, Tuscaloosa, Alabama
  - Cancer Treatment Services - AZ, Casa Grande, Arizona
  - Southwest Oncology Centers, Scottsdale, Arizona
  - Diablo Valley Oncology and Hematology Medical Group, Pleasant Hill, California
  - Parkridge Medical Center - Sara Cannon Cancer Center, Chattanooga, Tennessee

REFERENCES:
- [Background] Bhatnagar A, Loper A. The initial experience of electronic brachytherapy for the treatment of non-melanoma skin cancer. Radiat Oncol. 2010 Sep 28;5:87. doi: 10.1186/1748-717X-5-87. PMID 20875139